CLINICAL TRIAL: NCT02574663
Title: A Phase I Study Evaluating the Safety and Efficacy of TGR 1202 Alone and in Combination With Either Nab-paclitaxel + Gemcitabine or With FOLFOX in Patients With Select Relapsed or Refractory Solid Tumors
Brief Title: TGR-1202 Alone and in Combination With Either Nab-paclitaxel + Gemcitabine or With FOLFOX in Patients With Select Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-1202-102 (RM-404)
Record Dates: First submitted 2015-10-01; First posted 2015-10-14 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer; Colorectal Cancer; Rectal Cancer; Gastric Cancer; Esophageal Cancer; Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Gastrointestinal Stromal Tumors | interventions — umbralisib; 130-nm albumin-bound paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TGR-1202 (Experimental): TGR-1202 daily dose
  Interventions: Drug: TGR-1202
- TGR-1202 + nab-paclitaxel + gemcitabine (Experimental): TGR-1202 oral daily dose + nab-paclitaxel + gemcitabine both as an IV infusion
  Interventions: Drug: TGR-1202; Drug: nab-paclitaxel + gemcitabine
- TGR-1202 + FOLFOX (Experimental): TGR-1202 oral daily dose + oxaliplatin IV infusion + leucovorin IV infusion followed by 5-fluorouracil IV bolus followed by 5-FU IV infusion (FOLFOX regimen)
  Interventions: Drug: TGR-1202; Drug: Oxaliplatin + Folinic acid + Fluorouracil
- TGR-1202 + FOLFOX + Bevacizumab (Experimental): TGR-1202 oral daily dose + oxaliplatin IV infusion + leucovorin IV infusion followed by 5-fluorouracil IV bolus followed by 5-FU IV infusion (FOLFOX regimen) + bevacizumab IV infusion
  Interventions: Drug: TGR-1202; Drug: Oxaliplatin + Folinic acid + Fluorouracil + Bevacizumab

INTERVENTIONS:
Drug: TGR-1202 — TGR-1202 oral daily dose
Drug: nab-paclitaxel + gemcitabine — IV infusion
  Other Names: Abraxane (nab-paclitaxel) + Gemzar (gemcitabine)
  Arms: TGR-1202 + nab-paclitaxel + gemcitabine
Drug: Oxaliplatin + Folinic acid + Fluorouracil — IV infusion
  Other Names: Eloxatin (Oxaliplatin) + Leucovorin (Folinic acid) + 5-FU (Fluorouracil)
  Arms: TGR-1202 + FOLFOX
Drug: Oxaliplatin + Folinic acid + Fluorouracil + Bevacizumab — IV Infusion
  Other Names: Eloxatin (Oxaliplatin) + Leucovorin (Folinic acid) + 5-FU (Fluorouracil) + Avastin (Bevacizumab)
  Arms: TGR-1202 + FOLFOX + Bevacizumab

SUMMARY:
This is a Phase 1 multi-center study to assess the safety and efficacy of TGR-1202 as a single agent or in combination with nab-paclitaxel + gemcitabine or with FOLFOX in patients with select relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
TGR-1202 will be evaluated alone or in combination with nab-paclitaxel + gemcitabine or with FOLFOX in patients with adenocarcinoma of the pancreas, adenocarcinoma of the colon, rectum, gastric and GE junction cancer, and GI Stromal Tumor (GIST) who have relapsed from or are refractory to prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed:

  1. adenocarcinoma of the pancreas (pancreatic cancer)
  2. adenocarcinoma of the colon or rectum (colorectal cancer)
  3. adenocarcinoma of the gastric (gastric cancer)
  4. esophageal cancer
  5. gastrointestinal stromal tumor (GIST)
* Relapsed or refractory disease
* Measurable lesion by RECIST 1.1

Exclusion Criteria:

* Known Hepatitis B, C or HIV infection
* Previous therapy with any drug that inhibits the PI3K pathway
* Anti-tumor therapy within 21 days of study Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of safety and tolerability of TGR-1202 as a single agent and in combination in combination with nab-paclitaxel + gemcitabine, or with oxaliplatin + leucovorin + 5-FU (FOLFOX) or with FOLFOX + bevacizumab. | Up to 28 days after the last patient enrolled
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  Overall response rate with TGR-1202 as a single agent and in combination with nab-paclitaxel + gemcitabine, or with oxaliplatin + leucovorin + 5-FU (FOLFOX) or with FOLFOX + bevacizumab.
Duration of Response | Up to 1 year
  Duration of response with TGR-1202 as a single agent and in combination with nab-paclitaxel + gemcitabine, or with oxaliplatin + leucovorin + 5-FU (FOLFOX) or with FOLFOX + bevacizumab.
Pharmacokinetic (PK) profile of TGR-1202. Peak Plasma Concentration (Cmax). | At selected timepoints up through 6 months
  This endpoint will measure the plasma PK profile of TGR-1202 as a single agent and in combination with nab-paclitaxel + gemcitabine, or with oxaliplatin + leucovorin + 5-FU (FOLFOX) or with FOLFOX + bevacizumab.
Pharmacokinetic (PK) profile of TGR-1202. Time to Peak Plasma Concentration (Tmax). | At selected timepoints up through 6 months
Pharmacokinetic (PK) profile of TGR-1202. Area under the plasma concentration versus time curve (AUC) | At selected timepoints up through 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Study Chair — Sarah Cannon Research Instititue (SCRI)
Locations (1):
- TG Therapeutics Trial Site, Nashville, Tennessee, United States